CLINICAL TRIAL: NCT04489004
Title: Credit-AF: A Randomized Control Study of Driver Ablation Combined With Circumferential Pulmonary Vein Isolation Versus Stepwise Ablation as a Treatment in Patients With Persistent Atrial Fibrillation.
Brief Title: The Chinese Registration Study of Driver Ablation of Persistent Atrial Fibrillation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Credit-AF
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: Persistent Atrial Fibrillation; Driver ablation; Stepwise ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Driver ablation+CPVI (Experimental): Driver ablation plus CPVI (circumferential pulmonary vein isolation)
  Interventions: Procedure: Driver ablation+CPVI
- Stepwise ablation (Active Comparator): Stepwise ablation
  Interventions: Procedure: Stepwise ablation

INTERVENTIONS:
Procedure: Driver ablation+CPVI — Patients receive driver ablation and CPVI (circumferential pulmonary vein isolation).
  Arms: Driver ablation+CPVI
Procedure: Stepwise ablation — Patients receive stepwise ablation.
  Arms: Stepwise ablation

SUMMARY:
This is an open label, multi-center, randomized parallel control clinical trial, to demonstrate the role of driver mechanism in maintenance substrate of persistent atrial fibrillation, and evaluate the clinical outcomes of driver mapping and ablation strategy in patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
This is an open label, multi-center, randomized parallel control clinical trial. Patients with persistent atrial fibrillation are 1:1 randomized into the experimental group (driver ablation+ circumferential pulmonary vein isolation) or the control group (stepwise ablation). Postoperative atrial fibrillation recurrence rate and other indicators are analyzed to demonstrate the role of driver mechanism in maintenance substrate of persistent atrial fibrillation and evaluate the clinical outcomes of driver mapping and ablation strategy in patients with persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old;
2. Persistent AF;
3. nonresponse or intolerance to ≥1 antiarrhythmic drug. -

Exclusion Criteria:

1. With uncontrolled congestive heart failure;
2. Having significant valvular disease and/or prosthetic heart valve(s);
3. With myocardial infarction or stroke within 6 months of screening;
4. With Significant congenital heart disease;
5. Ejection fraction was <40% measured by echocardiography;
6. Allergic to contrast media;
7. Contraindication to anticoagulation medications;
8. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);
9. Left atrial (LA) thrombus measured by pre-procedure transesophageal echocardiography;
10. Having any contraindication to right or left sided heart catheterization;
11. Previous atrial fibrillation ablation;
12. Presence of an implanted cardioverter-defibrillator;
13. Any cardiac surgery within the past 2 months;
14. Poor general health;
15. Life expectancy less than 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1298 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation (AF) recurrence rate | up to 24 months after enrollment
  AF recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration.
Procedural AF termination rate | Before the end of procedure.
  AF termination is defined as conversion to sinus rhythm or a stable atrial flutter (AFL)/atrial tachycardia (AT).

SECONDARY OUTCOMES:
Postoperative atrial flutter (AFL) or atrial tachycardia (AT) rate | up to 24 months after enrollment
  Occurrence of AFL/AT is defined as presence of documented AFL/AT episodes of 30 seconds or longer duration.
Incidence of complications | up to 2 weeks after enrollment
  Complications include: death, atrioesophageal fistula, cardiac tamponade/perforation, myocardial infarction, stroke/cerebrovascular accident, thromboembolism, transient ischemic attack (TIA), diaphragmatic paralysis, pneumothorax, heart block, pulmonary vein stenosis, pulmonary edema, pericarditis, and major vascular access complication or bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China